# Effect Mindfulness Based Training on Attention, Hyperactivity and Emotion Regulation Among Children with ADHD: A Randomized Controlled Trails

| Contributing Authors: |
|---|
| Mohamed Hussein Atta *, |
| Lecturer, Psychiatric and Mental Health Nursing Department, Faculty of Nursing, Alexandria University, Egypt. ( <a href="mailto:mohamed-hussein@alexu.edu.eg">mohamed-hussein@alexu.edu.eg</a> ) |
| *Corresponding author ( <u>mohamed-hussein@alexu.edu.eg.</u> ) |
| Corresponding author at: Admeon Freemon st, Semoha, Alexandria, Egypt, Faculty of Nursing, Psychiatric Nursing Department, telephone +201067043760. |
| Abstract |
| Background: |
| The aim: |
| Setting: |
| Subjects |
| Tools: |
| Results: |
| Recommendation: |
| Keyword: |

#### Introduction

Attention-deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder that commonly affects children and adolescents and can persist into adulthood (Azzam et al., 2021; Liu et al., 2018). It is one of the leading causes for children to be referred to psychology and psychiatric clinics. A recent systematic review found that the global prevalence of ADHD is 7.6% (Salari et al., 2023), with higher estimates among children aged 3-17 years varying from 6% to 16% (Danielson et al., 2022). In Egypt, epidemiological studies indicate that ADHD is a widespread condition that affects 9.4 to 21.8% of children, which is higher than the worldwide incidence (Aboul-ata & Amin, 2015; Bishrry et al., 2018; EL-Gendy et al., 2017).

While research on the prevalence of ADHD in Egypt is limited, and further studies are needed to better understand the extent of this disorder in the country. Hence, implementing evidence-based practices to address the symptoms of ADHD is crucial to improving the well-being of both affected children and families (Aboul-ata & Amin, 2015; Bishrry et al., 2018; EL-Gendy et al., 2017).

ADHD symptoms can have a significant impact on the child and their family. The symptoms of hyperactivity, inattention, and impulsivity can affect the child's academic performance, social interactions, and overall quality of life. Children may struggle with tasks, organizing activities, and following instructions, and their emotions may be difficult to control. The family of a child with ADHD may also be affected, experiencing stress, frustration, and a sense of helplessness. This can lead to emotional exhaustion and financial strain for parents and caregivers due to the cost of treatment and missed work (Bishry et al., 2008; Peñuelas-Calvo et al. 2020)

Attention deficit is one of hallmark symptom of ADHD, making it difficult for them to concentrate, stay focused, and complete tasks. This can have a significant impact on their academic performance, social interactions, and self-esteem. In the classroom, children with ADHD may struggle with following instructions, organizing their work, and controlling their behavior. However, with proper support and intervention, children with ADHD can learn to manage their symptoms and lead successful lives (Bruno et al., 2023; Singh et al., 2015).

Moreover, hyperactivity is a common symptom of ADHD and can take various forms, such as fidgeting, restlessness, excessive talking, and impulsiveness. This can make it challenging for children to engage in calm activities, follow rules, and finish tasks. Additionally, they may find it difficult to socialize and maintain friendships as their behavior can be disruptive and overwhelming for others. The constant movement and restlessness can cause fatigue and difficulty sleeping, further affecting their daily life. This can be stressful for family members who may have difficulty managing the child's behavior and needs. However, with appropriate interventions and support, children with hyperactivity can learn to manage their symptoms and improve their overall well-being. (Hinshaw et al., 2021; Fioravante, Lozano-Lozano, Martella, 2022).

Emotion regulation is the ability to manage and control one's emotional responses to different environmental stimuli. Children diagnosed with (ADHD) often experience difficulties with emotion regulation. These challenges can take various forms, such as difficulty with emotional self-awareness and self-monitoring due to inattentive symptoms, impulsive emotional reactions due to impulsivity, and heightened emotional arousal and difficulty calming down due to hyperactivity (Soler-Gutiérrez, Pérez-González, & Mayas, 2023). These emotion regulation difficulties can have significant negative consequences for children with ADHD, including increased risk for anxiety and depression, social difficulties, and academic and occupational impairments (Walter et al., 2023). Therefore, it is crucial to address difficulties in emotion regulation, attention, and behavior as part of the comprehensive treatment of ADHD. Effective interventions, such as cognitive-behavioral therapy, mindfulness-based interventions, and medication management, can assist people with ADHD in developing effective emotion regulation skills and enhancing their overall functioning. (Haugan et al., 2022; Jenkins, et al., 2020; Lee, Chen & Lin, 2022).

Mindfulness training is a promising form of training for children with ADHD, as it focuses on attention and has gained empirical support as a complementary or alternative intervention. It involves increasing awareness and nonjudgmental observation of present-moment experiences while reducing automatic responding (Cairneross, & Miller 2016; Santonastaso et al., 2020). Attention regulation is a fundamental mechanism of mindfulness meditation, which involves training to sustain focus on present-moment experiences and gently shifting attention back to the meditation object when the mind drifts (Bishop, et al., 2004). Mindfulness meditation is a relatively new approach for reducing stress and emotion regulation difficulties among children. While researching the efficacy of mindfulness training in children is a new domain, existing evidence suggests that it has positive effects on psychological well-being, pain management, emotion dysregulation, negative behaviors, and cognitive/executive functions and attention (Evans et al., 2018; Zhang, Díaz-Román, & Cortese, 2018).

Nurses have an important role in caring for children with ADHD, particularly in the context of mindfulness-based interventions. They can provide education and support to both parents and children regarding the benefits of mindfulness practice and can help implement mindfulness programs in clinical and community settings. Nurses can assist children with ADHD to develop mindfulness skills, including paying attention to present-moment experiences and managing their emotions. This can be done through individual or group sessions, where nurses can guide children through various mindfulness exercises and provide feedback and support. Collaborating with other healthcare professionals such as psychologists and psychiatrists, nurses can ensure that children with ADHD receive comprehensive and coordinated care. By integrating mindfulness into their care approach, nurses can help enhance attention, emotion regulation, and overall well-being in children with ADHD.

| The research questi | ons: |
|---|---|
| | MATERIALS AND METHOD |
| MATERIALS | |
| I. Research de | esign: |
| II. Setting: | |
| III. Subjects: | |
| Tools: | |
| Four tools were used | for data collection in this study: |
| Tool I: A Socio-demographic and Academic Data Questionnaire: | |
| Part 1 Socio-demog<br>Part 2 Academic da<br>Tool III: | |
| Tool IV: | |
| Ethical approval and consent to participate. | |
| Declaration of Helsi<br>research ethics comm | carried out according to the relevant guidelines and regulations of the nki (DoH-Oct2008). Study procedures were revised and approved by the nittee of the faculty of nursing, Alexandria University and the Human Rights the of the General Secretariat of Mental Health, Ministry of Health, and |

## **Declaration**

The aim of the study is to:

Population in Cairo (IRB). An informed written consent was obtained from all patients after

explaining the purpose and nature of the study and who agreed to participate in the study.

## **Consent for publication**

Not applicable.

## Availability of data and materials

The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.

## **Competing interests**

No potential conflict of interest was reported by the authors.

## **Funding**

This research did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors.

#### **Authors contributions**

## Acknowledgements

Our sincere thanks go to all participants of the study.

### Reference

Aboul-ata, M. A., & Amin, F. A. (2015). The Prevalence of ADHD in Fayoum City (Egypt) Among School-Age Children: Depending on a DSM-5-Based Rating Scale. Journal of attention disorders, 22(2), 119-124. [https://doi.org/10.1177/1087054715576917

▶ (https://doi.org/10.1177/1087054715576917)

Azzam, H., Hasan, H., Elhabiby, M., El Ghamry, R., Mansour, M., & Elhamshary, M. (2021). Perceived parenting attitudes in relation to ADHD symptoms and aggressive behaviors in a sample of Egyptian children with ADHD. Middle East Current Psychiatry, 28(1), 18. [https://doi.org/10.1186/s43045-021-00055-7 ▶](https://doi.org/10.1186/s43045-021-00055-7)

Bishop, S. R., Lau, M., Shapiro, S., Carlson, L., Anderson, N., Carmody, J., Segal, Z., Abbey, S., Speca, M., Velting, D., et al. (2004). Mindfulness: A proposed operational definition. Clinical Psychology, 11, 230-241. doi: 10.1093/clipsy.bph077.

Bishry Z, Ramy HA, El-Shahawi HH, El-Sheikh MM, El-Missiry AA, El-Missiry MA (2018) Screening for ADHD in a sample of Egyptian adolescent school students. J Atten Disord 22(1):58–65

- Bruno, C., Havard, A., Gillies, M. B., Coghill, D., Brett, J., Guastella, A. J., Pearson, S.-A., & Zoega, H. (2023). Patterns of attention deficit hyperactivity disorder medicine use in the era of new non-stimulant medicines: A population-based study among Australian children and adults (2013-2020). Australian and New Zealand Journal of Psychiatry, 57(5), 675-685. doi: 10.1177/00048674221114782. PMID: 35999695.
- Cairncross, M., & Miller, C. J. (2016). The effectiveness of mindfulness-based therapies for ADHD: A meta-analytic review. Journal of Attention Disorders, 20(1), 1-17. doi: 10.1177/1087054713486512.
- Danielson ML, Holbrook JR, Newsome K., Charania SN, McCord RF, Kogan MD, Blumberg SJ. State-level estimates of the prevalence of parent-reported ADHD diagnosis and treatment among U.S. children and adolescents, 2016–2019. Journal of Attention Disorders, published online May 22, 2022.
- EL-Gendy SD, El-Bitar EA, El-Awady MA, Bayomy HE, Agwa EM. Attention-deficit/hyperactivity disorder: prevalence and risk factors in Egyptian primary school children. *The Egyptian Journal of Community Medicine*2017;35(1):1-16.
- Evans, S., Ling, M., Hill, B., Rinehart, N., Austin, D., & Sciberras, E. (2018). Systematic review of meditation-based interventions for children with ADHD. European Child & Adolescent Psychiatry, 27(1), 9-27. doi: 10.1007/s00787-017-1024-6.
- Fioravante, I., Lozano-Lozano, J. A., & Martella, D. (2022). Attention deficit hyperactivity disorder: A pilot study for symptom assessment and diagnosis in children in Chile. Frontiers in Psychology, 13, 946273. doi: 10.3389/fpsyg.2022.946273.
- Haugan, A. L. J., Sund, A. M., Young, S., Thomsen, P. H., Lydersen, S., & Nøvik, T. S. (2022). Cognitive behavioural group therapy as addition to psychoeducation and pharmacological treatment for adolescents with ADHD symptoms and related impairments: A randomised controlled trial. BMC Psychiatry, 22, 375. doi: 10.1186/s12888-022-04019-6. PMID: 35655149. PMCID: PMC9164353.
- Hinshaw, S. P., Nguyen, P. T., O'Grady, S. M., & Rosenthal, E. A. (2021). Annual Research Review: Attention-deficit/hyperactivity disorder in girls and women: underrepresentation, longitudinal processes, and key directions. Journal of Child Psychology and Psychiatry, 62(8), 885-908. doi: 10.1111/jcpp.13359.
- Jenkins, R., Othieno, C., Okeyo, S., Aruwa, J., Wallcraft, J., Jenkins, B., & Bassett, P. (2020). Health system challenges and solutions for better management of child and adolescent mental health in low-income and middle-income countries. AIMS Public Health, 7(1), 93-109. doi: 10.3934/publichealth.2020009.

Liu A, Xu Y, Yan Q, Tong L. The prevalence of attention deficit/hyperactivity disorder among chinese children and adolescents. Sci Rep. 2018;8(1):1–15.

Overall, ADHD is a significant public health concern worldwide, and it is important to continue researching its prevalence and impact on children's development. Early diagnosis and intervention are crucial to improving outcomes for children with ADHD and helping them reach their full potential.

Peñuelas-Calvo, I., Palomar-Ciria, N., Porras-Segovia, A., Miguélez-Fernández, C., Baltasar-Tello, I., Perez-Colmena, S., Delgado-Gómez, D., Carballo, J. J., & Baca-García, E. (2020). Impact of ADHD symptoms on family functioning, family burden and parents' quality of life in a hospital area in Spain. Revista de Psiquiatría y Salud Mental, 35(3), 166-172. doi: 10.1016/j.rpsm.2019.11.002

Salari, N., Ghasemi, H., Abdoli, N., Rahmani, A., Shiri, M. H., Hashemian, A. H., Akbari, H., & Mohammadi, M. (2023). The global prevalence of ADHD in children and adolescents: A systematic review and meta-analysis. Italian Journal of Pediatrics, 49(1), 48. [https://doi.org/10.1186/s13052-023-01190-1]/[https://doi.org/10.1186/s13052-023-01190-1]

Santonastaso, O., Zaccari, V., Crescentini, C., Fabbro, F., Capurso, V., Vicari, S., & Menghini, D. (2020). Clinical application of mindfulness-oriented meditation: A preliminary study in children with ADHD. International Journal of Environmental Research and Public Health, 17(18), 6916. doi: 10.3390/ijerph17186916.

Singh, A., Yeh, C. J., Verma, N., & Das, A. K. (2015). Overview of attention deficit hyperactivity disorder in young children. Health Psychology Research, 3(2), 2115. doi: 10.4081/hpr.2015.2115. PMID: 26973960. PMCID: PMC4768532.

Soler-Gutiérrez, A. M., Pérez-González, J. C., & Mayas, J. (2023). Evidence of emotion dysregulation as a core symptom of adult ADHD: A systematic review. PLoS One, 18(1), e0280131. doi: 10.1371/journal.pone.0280131.

Walter, A., Martz, E., Weibel, S., & Weiner, L. (2023). Tackling emotional processing in adults with attention deficit hyperactivity disorder and attention deficit hyperactivity disorder + autism spectrum disorder using emotional and action verbal fluency tasks. Frontiers in Psychiatry, 14, 1098210. doi: 10.3389/fpsyt.2023.1098210.

- Zhang, J., Díaz-Román, A., & Cortese, S. (2018). Meditation-based therapies for attention-deficit/hyperactivity disorder in children, adolescents, and adults: A systematic review and meta-analysis. Evidence-Based Mental Health, 21, 87-94. doi: 10.1136/ebmental-2018-300022.
- Lee, Y.-C., Chen, C.-R., & Lin, K.-C. (2022). Effects of mindfulness-based interventions in children and adolescents with ADHD: A systematic review and meta-analysis of randomized

controlled trials. International Journal of Environmental Research and Public Health, 19(22), 15198. doi: 10.3390/ijerph192215198. PMID: 36429915. PMCID: PMC9690476.